CLINICAL TRIAL: NCT03972033
Title: Multicenter RCT Comparing EMDR and CBT Efficacy for Treatmen of Resistant Depression
Brief Title: RCT Comparing EMDR and CBT for Treatment of Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: EMDR Europe (Industry)
Responsible Party: Principal Investigator, luca ostacoli, Full Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMDRvsCBT
Record Dates: First submitted 2019-03-27; First posted 2019-06-03 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Eye Movement Desensitization and Reprocessing; Cognitive Behavioral Therapy; Neurobiological Processing; Depression; Functional Magnetic Resonance Imaging; High Definition Electroencefalography; Heart Rate Variability
Keywords: depression; neurobiology of emotions; Cognitive Behavioral Therapy; Eye Movement Desensitization and Reprocessing; trauma; psychotherapy
MeSH Terms: conditions — Depression; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The design of the study is a randomized controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors doesn't know the patient group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing (Experimental): The DeprEND manualized protocol (Hofmann, Ostacoli, et al., 2015) is based on the eight-phase protocol by Shapiro (2001) that was adapted for the treatment of depression by the European Depression EMDR Network and used in previous studies (Hase et al., 2015; Hofmann et al., 2014; Ostacoli et al., 2018). EMDR targets will be selected using the Adaptive Information Processing model that looks for stressful events linked with depression. The DeprEnd Fidelity Rating Scale will be used to assess treatment fidelity. The scale will be completed by trained EMDR therapists who will listen to the audio recordings of the sessions.
  In each centre, EMDR is provided by psychotherapists specialized in Level II EMDR and with a minimum of three years of experience in treating patients with depression. They receive extensive training and supervision in the manualized protocol established for the study, from a certified senior EMDR instructor.
  Interventions: Behavioral: EMDR
- Cognitive Behavioral Therapy (Active Comparator): Treatment protocol is based on the principles described by Beck (Beck et al., 1979) will be utilized. The treatment includes behavioral activation and cognitive restructuring with homework assignments. In each centre, CBT treatment is performed by psychotherapists with certified training in CBT techniques and a minimum of three years of experience in treating patients with depression. They receive regular CBT supervision to ensure that the quality of their CBT treatment was maintained.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: EMDR — Treatments will be independent and blinded to the clinical psychologists conducting the clinical assessments. EMDR and CBT treatments will be provided for 16 weeks, each comprising 16 weekly individual sessions. Interventions will be conducted according to published treatment manuals. All treatment sessions will be video recorded for fidelity rating and supervision.
  As a safety criterion, if severe worsening of symptoms is observed, patients are withdrawn from their assigned treatment arm.
  Other Names: Eye Movement Desensitization and Reprocessing
  Arms: Eye Movement Desensitization and Reprocessing
Behavioral: CBT — Treatments will be independent and blinded to the clinical psychologists conducting the clinical assessments. EMDR and CBT treatments will be provided for 16 weeks, each comprising 16 weekly individual sessions. Interventions will be conducted according to published treatment manuals. All treatment sessions will be video recorded for fidelity rating and supervision.
  As a safety criterion, if severe worsening of symptoms is observed, patients are withdrawn from their assigned treatment arm.
  Other Names: Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Depression is one of the most common invalidating mental disorders, ranked by World Health Organization as the single largest contributor to global disability. Current recommended treatments for depression include antidepressant medication and according to guidelines, Cognitive Behavioral Therapy (CBT) and Interpersonal Therapy (IPT). Despite encouraging preliminary results (e.g., Matthijssen et al., 2020), Eye Movement Desensitization and Reprocessing (EMDR) therapy is not yet recognized as an effective therapy for depression by APA and NICE. The project aims to conduct a large multisite study that addresses the shortcomings of previous efficacy research on EMDR for depression. The primary aim is to evaluate the effectiveness of EMDR therapy in reducing depressive symptoms in adults with major depression as compared to CBT. Secondary aims of the study are the effectiveness of EMDR, as compared to CBT and TAU, in improving anxiety, and other symptoms. It is hypothesized that EMDR is not inferior to CBT.

DETAILED DESCRIPTION:
The study is a multicenter clinical randomized controlled trial, conducted in Italy, USA and UK that will assess the effectiveness of EMDR therapy compared to CBT and TAU. Patients will be recruited at four clinical centers: Turin and Rome in Italy, and Kansas City in USA. The study protocol was approved by the local research ethics committee in each of the countries where the intervention is implemented.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of Major Depressive Disorder, single episode or recurrent, according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
2. a score of at least 20 on Beck's Depression Inventory-II (BDI-II);
3. having received ADM treatment with a stable dose for at least six weeks and maintained stable during treatment;
4. legal capacity to consent to the treatment.

Exclusion Criteria:

1. diagnosis of current PTSD (assessed with MINI-Plus and the International Trauma Questionnaire - ITQ, Cloitre et al., 2018);
2. diagnosis of complex PTSD (assessed with the ITQ);
3. history of psychotic symptoms or schizophrenia;
4. bipolar disorder or dementia;
5. cluster A and B severe personality disorders;
6. dissociative symptoms (DES-B score >2);
7. any substance-related abuse or dependence disorder (except those involving nicotine) in the 6 months prior to the study;
8. a serious, unstable medical condition;
9. a severely unstable social and economic condition (e.g. no fixed abode; job loss without any other source of income);
10. being pregnant;
11. acute suicidality that needs hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup).
  Beck Depression Inventory II (BDI-II)
changes in depressive symptoms | week 0, week 16, week 40
  Hamilton Depression Rating Scale (HDRS)
changes in cognitive component of depressive syndrome | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Beck Hopelessness Scale (BHS)
changes in HD-EEG | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  HD-EEG in resting state phase and a second phase with a task
changes in fMRI | month 0 (T0)
  fMRI in resting state phase and a second phase with a task
changes in HRV | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  HRV detection during hdEEG assessment
psychiatric diagnosis | month 0 (T0)
  Structured Clinical Interview for DSM-5 (SCID-5)
changing in depressive symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup) and every week
  Patient Health Questionnaire-9 (PHQ-9)

SECONDARY OUTCOMES:
addressing potentially traumatizing events | month 0 (T0)
  Traumatic Experience Checklist (TEC)
assessing childhood trauma | month 0 (T0)
  Childhood Trauma Questionnaire (CTQ)
evaluating the quality of relationships | month 0 (T0)
  Relationship Questionnaire (RQ)
changing in dissociative symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Brief Dissociative Experiences Scale (DES-B)
changing in autonomic symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Composite Autonomic Symptom Score (COMPASS-31)
changing in the emotional regulation | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Difficulties in Emotion Regulation Scale (DERS)
changing in the dimensions of the emotional style | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Emotional Style Questionnaire (ESQ)
changing in quality of sleep, in particular insomnia | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Insomnia Severity Index (ISI)
changing in physical activity habits | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  International Physical Activity Questionnaire Short Form (IPAQ-SF)
changing in post-traumatic symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  International Trauma Questionnaire
changing in suicidal thinking | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Paykel Suicide Scale
changing in stress | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  Perceived Stress Scale (PSS)
changing in post-traumatic stress symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup)
  PTSD Checklist for DSM-5 (PCL-5)
assessing disability and functional impairment as a result of treatment | 1 month time frame
  Sheehan Disability Scale for Treatment Induced Impairment (SDS-T)
changing in anxiety symptoms | month 0 (T0, baseline), month 4 (T1, post-treatment), month 10 (T2, followup), month 22 (T3, followup) and every week
  General Anxiety Disorder-7 (GAD-7)

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided